CLINICAL TRIAL: NCT00357409
Title: GABA Levels in the Occipital Cortex of Blind Human Subjects
Brief Title: GABA Levels in the Brains of Blind People
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020124; 02-N-0124
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-03-03

CONDITIONS: Vision; Blind
Keywords: GABA; Occipital; Vision; Plasticity; MRS; Blind

SUMMARY:
In blind individuals, the occipital cortex becomes capable of processing tactile and auditory information, a phenomenon described as crossmodal plasticity. GABA is the major inhibitory neurotransmitter in the brain and a possible candidate to mediate this form of human plasticity. We intend to use magnetic resonance spectroscopy (MRS) to measure GABA and hypothesize that GABA levels in the occipital cortex of blind humans will be lower than in sighted controls. Such decrease could possibly mediate compensatory changes in the occipital cortex of the blind.

Objective

Early blind subjects exhibit better tactile acuity than late blinds or sighted individuals. The purpose of the study is the determine GABA levels in the human occipital cortex after long-term light deprivation (blindness).

Study Population

Our experiments will make use of early blind, late blind, and sighted control subjects.

Design

Subject will be identified and will receive clinical and neurological examinations at the NIH. MRS studies will be performed at NIH MRI Center with 3Tesla Magnet. Each subject head will be positioned in an adjustable holder (designed for minimal motion and maximal comfort) such that a flat coil lay just below the occipital cortex. The sequence has been described before [33]. The individuals who perform the data analysis will be blind to the purpose of the experiments.

Outcome measures

The concentration of GABA from the 14 ml voxel over the visual cortex will be measured. Edited proton spectrum of GABA will be compared with the edited sub spectrum of creatine for a concentration reference.

DETAILED DESCRIPTION:
In blind individuals, the occipital cortex becomes capable of processing tactile and auditory information, a phenomenon described as crossmodal plasticity. GABA is the major inhibitory neurotransmitter in the brain and a possible candidate to mediate this form of human plasticity. We intend to use magnetic resonance spectroscopy (MRS) to measure GABA and hypothesize that GABA levels in the occipital cortex of blind humans will be lower than in sighted controls. Such decrease could possibly mediate compensatory changes in the occipital cortex of the blind.

Objective

Early blind subjects exhibit better tactile acuity than late blinds or sighted individuals. The purpose of the study is the determine GABA levels in the human occipital cortex after long-term light deprivation (blindness).

Study Population

Our experiments will make use of early blind, late blind, and sighted control subjects.

Design

Subjects will be identified and will receive clinical and neurological examinations at the NIH. MRS studies will be performed at NIH MRI Center with 3Tesla Magnet. Each subject head will be positioned in an adjustable holder (designed for minimal motion and maximal comfort) such that a flat coil lay just below the occipital cortex. The sequence has been described before. The individuals who perform the data analysis will be blind to the purpose of the experiments.

Outcome measures

The concentration of GABA from the 14 ml voxel over the visual cortex will be measured. Edited proton spectrum of GABA will be compared with the edited sub spectrum of creatine for a concentration reference.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must be between 18 and 55 years of age.

Healthy sighted volunteers. Legally blind subjects with blindness secondary to retinal lesions or eye removal acquired at ages earlier than 4 years old (EARLY) and after 13 years of age (LATE). The rationale for the distinction is based in our previous studies that indicate different magnitude of brain plasticity depending on the age of acquisition of blindness.

EXCLUSION CRITERIA:

Exclusion criteria will be those of MRI procedures:

Pregnant women tested after urine pregnancy test.

Subjects with metal in the cranium except mouth.

Subjects with metal fragments from occupational exposure or surgical clips in or near the brain.

Subjects with blood vessel, cochlear or eye implants.

Subjects with increased intracranial pressure as evaluated by clinical means.

Subjects with cardiac or neural pacemakers.

Subjects with intracardiac lines and implanted medication pumps.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39
Dates: Start 2002-02-11; Study Completion 2008-03-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Micheva KD, Beaulieu C. Neonatal sensory deprivation induces selective changes in the quantitative distribution of GABA-immunoreactive neurons in the rat barrel field cortex. J Comp Neurol. 1995 Oct 30;361(4):574-84. doi: 10.1002/cne.903610403. PMID 8576415